CLINICAL TRIAL: NCT04281654
Title: Effects of Arts Engagement Programs on Physical Performance, Cognition, Social Isolation, and Self Perception in Older Adults
Brief Title: Effects of Arts Engagement on Physical Performance, Cognition, Social Isolation, and Self-Perception in Older Adults
Acronym: SHARe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Collaborators: National Endowment for the Arts, United States (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1428455-1
Record Dates: First submitted 2019-07-29; First posted 2020-02-24 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Social Isolation; Mental Status Change; Cognitive Impairment; Physical Activity; Quality of Life; Self-Perception
Keywords: Dance; Music; Social Conversation
MeSH Terms: conditions — Social Isolation; Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ballroom Dance (Experimental): The Dance group participants will take part in ballroom dance lessons twice/week for 45-minutes/session for 10 weeks
  Interventions: Other: Active Social Conversation
- Ukulele (Experimental): The Music group participants will take part in ukulele lessons twice/week for 45-minutes/session for 10 weeks
  Interventions: Other: Active Social Conversation
- Control (Active Comparator): The Control group participants will meet 2 times per week for 45-minutes/session for 10 weeks to participate in a social conversational group for 10 weeks
  Interventions: Other: Active Social Conversation

INTERVENTIONS:
Other: Active Social Conversation — Active Social Conversation
  Other Names: Active Control

SUMMARY:
The purpose of this community-engaged project is to examine how taking part in different arts (dance & music), compared to control (no arts) affects older adults' Health-Related Quality of Life (HRQoL using the Short Form-20(SF) form), physical performance (Short Physical Performance Battery-SPPB), cognition (using the Montreal Cognitive Assessment-MoCA), social engagement (National Social Life, Health, & Aging Project-NSHAP survey), and perceptions of self (focus interviews).

DETAILED DESCRIPTION:
In this Randomized-Controlled-Trial, 60 adults (20/condition) will take part in 20, 45-minute sessions (ballroom dance, ukulele/guitar playing, or control- i.e. social conversation), 2 times/week for 10 weeks.

While the investigators know that arts participation improves function in older adults, exact effects of different arts programs on health outcomes remains unclear.

The investigators plan to fill this gap by studying how different arts participation affect health outcomes.

The overall aim is to study how arts engagement helps older adults remain active and influences physical, psychological, and emotional functioning.

ELIGIBILITY:
Inclusion Criteria:

* Be healthy,
* > 65 years of age and able to take part in learning music, or ballroom dance.

Exclusion Criteria:

* Presence of a co-morbid mental health diagnosis or other physical or behavioral challenges that the study staff assess as rendering the participant unable or unsafe to participate in the study.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2020-04-26 (Actual)

PRIMARY OUTCOMES:
Change in Physical Performance using the Short Physical Performance Battery (SPPB) | Pre (Week 0), Post 1 (Week 10) and Post 2 (Week 15) Intervention
  The Short Physical Performance Battery (SPPB) is an assessment tool for evaluation of lower extremity functioning in older persons. In this tool, participants will perform the 3 SPPB components: 1) Ability to stand for 10 sec with feet in 3 different positions (together side-by-side, semi-tandem, and tandem), 2) Two timed trials of a 4-m walk (fastest recorded), and 3) Time to rise from a chair five times. The subtests are scored from 0-4. The overall SPPB is scored from 0 (Minimum) to 12 (Maximum score) with higher scores indicating better lower extremity function.

SECONDARY OUTCOMES:
Change in Cognition using Montreal Cognitive Assessment (MOCA) survey | Pre (Week 0), Post 1 (Week 10) and Post 2 (Week 15) Intervention
  The Montreal Cognition Assessment (MoCA) is a brief, 30-question test designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. MoCA scores range between 0-30. A score of 26 or over is considered normal.
Change in Self-Perception Post Intervention Focus Interview | Post 1 (Week 10) and Post 2 (Week 15) Intervention
  In these interviews participants discuss how they self-perceive any physical, mental, and social changes they underwent as a result of taking part in the interventions
Change in Social Connections using the Social Connections Survey | Post 1 (Week 10) and Post 2 (Week 15) Intervention
  Participants complete questions from the National Social Life, Health, and Aging Project (NSHAP) measure perceived social connection and isolation. These questions ask participants about 1) Support from partner (we are using 3 of the 6 questions); 2) Support from family (we are using 3 of the 5 questions); 3) Support from friends (we are using 3 of the 5 questions). All questions are on a 4-point frequency range from "never" to "often", except for 2 questions. Question #1 construct one is on a 7-point scale from "very unhappy to "very happy" and question #5 construct two is on a 6-point scale from "none" to "more than 20". The 7 items with the same frequency anchors will be summed; the other two items will be analyzed as one-item indicators.

CONTACTS AND LOCATIONS:
Overall Officials: Jatin P Ambegaonkar, PhD, Principal Investigator — George Mason University
Locations (1):
- Hylton Performing Arts Center, Manassas, Virginia, United States

IPD SHARING:
Plan to Share IPD: No